CLINICAL TRIAL: NCT01574716
Title: A Study of the Safety and Efficacy of the Combination of Gemcitabine and Docetaxel With MORAb-004 in Metastatic Soft Tissue Sarcoma
Brief Title: Sarcoma Study of MORAb-004 Utilization: Research and Clinical Evaluation
Acronym: SOURCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MORAb-004-203-STS; 2012-001399-12 (EudraCT Number)
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2016-11

CONDITIONS: Metastatic Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — ontuxizumab; Gemcitabine; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MORAb-004, gemcitabine, docetaxel (Experimental)
  Interventions: Drug: MORAb-004; Drug: Gemcitabine; Drug: Docetaxel
- Placebo, gemcitabine, docetaxel (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Placebo

INTERVENTIONS:
Drug: MORAb-004 — IV, Days 1 and 8 of every cycle until disease progression
  Arms: MORAb-004, gemcitabine, docetaxel
Drug: Gemcitabine — IV, Days 1 and 8 of each cycle until disease progression
  Arms: MORAb-004, gemcitabine, docetaxel
Drug: Docetaxel — IV, Day 8 of every cycle until disease progression
  Arms: MORAb-004, gemcitabine, docetaxel
Drug: Gemcitabine — IV, Days 1 and 8 of each cycle until disease progression
  Arms: Placebo, gemcitabine, docetaxel
Drug: Docetaxel — IV, Day 8 of every cycle until disease progression
  Arms: Placebo, gemcitabine, docetaxel
Drug: Placebo
  Arms: Placebo, gemcitabine, docetaxel

SUMMARY:
This study is being done to see if MORAb-004 increases the effectiveness of the chemotherapies gemcitabine and docetaxel in people with metastatic Soft Tissue Sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Be surgically sterile or consent to use a medically acceptable method of contraception throughout the study period
* Have a histologically confirmed diagnosis of mSTS as defined by the 4 specified study subgrouped
* Have been treated in the metastatic setting with 0 to 2 prior systemic regimens for mSTS (Systemic treatment regimens given in the neoadjuvant setting and maintenance therapies will not be considered as regimens in the metastatic setting for the purposes of this protocol. Prior anthracycline-based regimen is allowable but not required. Subjects with extra-skeletal small round blue cell sarcomas, including rhabdomyosarcomas, must have exhausted or be intolerant of standard first line anthracycline-based chemotherapy.)
* Have measurable disease, as defined by RECIST v 1.1 assess within 2 weeks of study entry and have radiologically documented disease progression greater than or equal to a 10% increase in the sum of the longest diameters of target lesions present within 6 months prior to randomization
* Have tumor tissue available for TEM-1 biomarker studies
* Be willing and able to provide written informed consent

Exclusion Criteria:

* Have received more than 2 prior systemic treatment regimens for mSTS
* Have received either gemcitabine or docetaxel in any previous treatment for mSTS (regardless of the line of treatment)
* Have a diagnosis of primary bone sarcoma of any histological type.
* Have a history of clinically significant heart disease, or clinically significant arrhythmia on ECG within the past 6 months
* Have a history of allergic reaction to prior monoclonal antibody or biologic agent
* Have received previous treatment with MORAb-004 (anti-TEM-1)
* Have a medical condition with a high risk of bleeding (e.g., a known bleeding disorder, a coagulopathy, or a tumor that involves the major vessels) or have a recent (within past 6 months) history of a significant bleeding event
* Have undergone major surgical procedures or open biopsy, have significant traumatic injury within 30 days prior to the first date of study treatment, or have major surgical procedures anticipated during the study
* Have a serious non-healing wound, an ulcer (including gastrointestinal), or a bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2015-08-11 (Actual); Study Completion 2016-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (19):
  - Sarcoma Oncology Center, Santa Monica, California
  - UCLA, Santa Monica, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Mayo Clinic - Rochester, Rochester, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Seattle Care Alliance, Seattle, Washington
- Australia (5):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- UZ Leuven Medical Oncology, Leuven, Belgium
- France (2):
  - Institut Gustave Roussy, Villejuif
  - University of Claude Bernard, Villeurbanne
- Istituto Ortopedico Rizzoli, Bologna, Italy
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Jones RL, Chawla SP, Attia S, Schoffski P, Gelderblom H, Chmielowski B, Le Cesne A, Van Tine BA, Trent JC, Patel S, Wagner AJ, Chugh R, Heyburn JW, Weil SC, Wang W, Viele K, Maki RG. A phase 1 and randomized controlled phase 2 trial of the safety and efficacy of the combination of gemcitabine and docetaxel with ontuxizumab (MORAb-004) in metastatic soft-tissue sarcomas. Cancer. 2019 Jul 15;125(14):2445-2454. doi: 10.1002/cncr.32084. Epub 2019 Apr 29. PMID 31034598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 31 investigative sites in the United States, Australia, Italy, Netherlands, France and Belgium from 07 August 2012 to 02 August 2016.
Pre-assignment Details: In Part 1, a total of 16 participants were enrolled and treated in the study. A total of 225 participants were screened for entry into Part 2 of the study. Of these 225 participants, 46 were screen failures and 209 were randomized into the study, of which 207 participants were treated.
Groups:
- Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel: Participants received MORAb-004 4 milligram per kilogram (mg/kg), infusion, intravenously on Days 1 and 8 in combination with gemcitabine 900 milligram per square meter (mg/m^2), infusion, intravenously on Days 1 and 8 and docetaxel, infusion, intravenously on Day 8 of each 21-day treatment cycle until disease progression (approximately 28 cycles). MORAb-004 was administered after the administration of gemcitabine on Day 1 and after the administration of gemcitabine/docetaxel on Day 8 in each 21-day treatment cycle.
- Part 1: MORAb-004 6.0 mg/kg + Gemcitabine/Docetaxel: Participants received MORAb-004 6 mg/kg, infusion, intravenously on Days 1 and 8 in combination with gemcitabine 900 mg/m^2, infusion, intravenously on Days 1 and 8 and docetaxel 75 mg/m^2, infusion, intravenously on Day 8 of each 21-day treatment cycle until disease progression (approximately 28 cycles). MORAb-004 was administered after the administration of gemcitabine on Day 1 and after the administration of gemcitabine/docetaxel on Day 8 in each 21-day treatment cycle.
- Part 1: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel: Participants received MORAb-004 8 mg/kg, infusion, intravenously on Days 1 and 8 in combination with gemcitabine 900 mg/m^2, infusion, intravenously on Days 1 and 8 and docetaxel 75 mg/m^2, infusion, intravenously on Day 8 of each 21-day treatment cycle until disease progression (approximately 28 cycles). MORAb-004 was administered after the administration of gemcitabine on Day 1 and after the administration of gemcitabine/docetaxel on Day 8 in each 21-day treatment cycle.
- Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel: Participants received MORAb-004 8.0 mg/kg, infusion, intravenously on Days 1 and 8 in combination with gemcitabine 900 mg/m^2, infusion, intravenously on Days 1 and 8 and docetaxel 75 mg/m^2, infusion, intravenously on Day 8 of each 21-day treatment cycle for until disease progression (approximately 31 cycles). MORAb-004 was administered after the administration of gemcitabine on Day 1 and after the administration of gemcitabine/docetaxel on Day 8 in each 21-day treatment cycle.
- Part 2: Placebo + Gemcitabine/Docetaxel: Participants received normal saline (0.9 percent [%] sodium chloride), infusion, intravenously on Days 1 and 8 in combination with gemcitabine 900 mg/m^2, infusion, intravenously on Days 1 and 8 and docetaxel 75 mg/m^2, infusion, intravenously on Day 8 of each 21-day treatment cycle for until disease progression (approximately 31 cycles). Normal saline (0.9% sodium chloride) was administered after the administration of gemcitabine on Day 1 and after the administration of gemcitabine/docetaxel on Day 8 in each 21-day treatment cycle.
Period: Part 1
Arm/Group | Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 6.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Started | 3 | 4 | 9 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 9 | 0 | 0
Not completed — Death | 3 | 1 | 8 | 0 | 0
Not completed — Discontinuation of study by sponsor | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 6.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Started | 0 | 0 | 0 | 139 | 70
Treated Participants (MORAb: 2 discontinued prior to treatment. Placebo: 3 randomized but received MORAb are in MORAb.) | 0 | 0 | 0 | 140 | 67
Completed | 0 | 0 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 137 | 70
Not completed — Progressive disease | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 76 | 35
Not completed — Discontinuation of study by sponsor | 0 | 0 | 0 | 51 | 31
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 4
Not completed — Brain metastases | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Part 1: The intent-to-treat (ITT)/Safety population (SP) included all treated participants and was analyzed by treatment dose level. Part 2: The ITT population consisted of all randomized participants and were analyzed according to the treatment assigned by the interactive randomization system (IxRS).
Groups:
- Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel: Participants received MORAb-004 4 mg/kg, infusion, intravenously on Days 1 and 8 in combination with gemcitabine 900 mg/m^2, infusion, intravenously on Days 1 and 8 and docetaxel, infusion, intravenously on Day 8 of each 21-day treatment cycle until disease progression (approximately 28 cycles). MORAb-004 was administered after the administration of gemcitabine on Day 1 and after the administration of gemcitabine/docetaxel on Day 8 in each 21-day treatment cycle.
- Part 2: Placebo + Gemcitabine/Docetaxel: Participants received normal saline (0.9% sodium chloride), infusion, intravenously on Days 1 and 8 in combination with gemcitabine 900 mg/m^2, infusion, intravenously on Days 1 and 8 and docetaxel 75 mg/m^2, infusion, intravenously on Day 8 of each 21-day treatment cycle for until disease progression (approximately 31 cycles). Normal saline (0.9% sodium chloride) was administered after the administration of gemcitabine on Day 1 and after the administration of gemcitabine/docetaxel on Day 8 in each 21-day treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 6.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel | Total
Number analyzed (Participants) | 3 | 4 | 9 | 139 | 70 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 8 | 103 | 49 | 166
  >=65 years | 0 | 1 | 1 | 36 | 21 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 63 | 32 | 102
  Male | 1 | 2 | 6 | 76 | 38 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 18 | 8 | 29
  Not Hispanic or Latino | 2 | 4 | 7 | 119 | 61 | 193
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 3 | 8 | 116 | 57 | 185
  Black or African American | 1 | 1 | 0 | 12 | 9 | 23
  Asian | 1 | 0 | 1 | 7 | 2 | 11
  Chinese | 0 | 0 | 0 | 0 | 2 | 2
  American Indian or Alaskan Native | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Radiologic Progression-free Survival (PFS)
Description: PFS was defined as the time (in weeks) from the date of randomization to the date of first observation of disease progression according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or date of death, regardless of the cause.
Time Frame: From date of first dose until date of first observation of disease progression, or death due to any cause (up to approximately 3 years)
Population: The ITT population consisted of all randomized participants and were analyzed according to the treatment assigned by the IxRS.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Number analyzed (Participants) | 139 | 70
weeks | 18.7 [11.6 to 27.4] | 24.1 [11.1 to 36.1]
Statistical Analysis 1: Comparison: Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel vs Part 2: Placebo + Gemcitabine/Docetaxel; Test type: Superiority; p = 0.6562, Log Rank; Two-sided log-rank test; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.77 to 1.50] — Based on Cox PH model

2. Secondary Outcome: Part 2: Symptomatic Progression-free Survival
Description: PFS including symptomatic progression was defined as the time (in weeks) from the date of randomization to the date of the first observation of disease progression according to RECIST 1.1, symptomatic progression, or death due to any cause.
Time Frame: From date of first dose until date of first observation of disease progression, symptomatic progression, or death due to any cause (up to approximately 3 years)
Population: The ITT population consisted of all randomized participants and were analyzed according to treatment assigned by the IxRS.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Number analyzed (Participants) | 139 | 70
weeks | 18.1 [11.3 to 24.0] | 24.0 [10.7 to 36.1]
Statistical Analysis 1: Comparison: Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel vs Part 2: Placebo + Gemcitabine/Docetaxel; Test type: Superiority; p = 0.4469, Log Rank; Two-sided log-rank test; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.82 to 1.57] — Based on Cox PH model

3. Secondary Outcome: Part 2: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of randomization to the date of death, regardless of the cause.
Time Frame: From date of first dose until date of death from any cause (up to approximately 3.5 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Number analyzed (Participants) | 139 | 70
months | 18.3 [16.2 to 21.1] | 21.1 [14.2 to NA] — The upper limit of confidence interval (CI), was not estimable since high number of participants were censored from analysis.
Statistical Analysis 1: Comparison: Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel vs Part 2: Placebo + Gemcitabine/Docetaxel; Test type: Superiority; p = 0.3153, Log Rank; Two-sided log-rank test; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.82 to 1.83] — Based on Cox PH model

4. Secondary Outcome: Part 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of subjects with either a complete response (CR) or a partial response (PR) based on RECIST 1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR was defined as at least a 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first dose until disease progression (up to approximately 3.5 years)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Number analyzed (Participants) | 139 | 70
percentage of participants | 19.4 | 20.0
Statistical Analysis 1: Comparison: Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel vs Part 2: Placebo + Gemcitabine/Docetaxel; Difference equal to (=) (MORAb 8.0 mg/kg + Gemcitabine/Docetaxel) minus (Placebo + Gemcitabine/Docetaxel). Confidence interval based on a normal approximation to the binomial distribution; Test type: Superiority; p = 1.000, Log Rank; Two-sided log-rank test; Difference = -0.6, 95% CI 2-sided [-12.0 to 10.9] — Based on Cox PH model

5. Secondary Outcome: Part 2: Radiologic Progression-free Survival Rate (PFR)
Description: Radiologic progression-free survival rate was defined as the percentage of subjects achieving radiologic PFS at the pre-specified time points.
Time Frame: Weeks 12, 24, 48 and 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Number analyzed (Participants) | 139 | 70
percentage of participants
  12 weeks | 57.6 | 61.8
  24 weeks | 43.3 | 51.0
  48 weeks | 24.5 | 25.2
  52 weeks | 20.8 | 21.4

6. Secondary Outcome: Part 2: Number of Participants Who Had Relationship Between MORAb-004 Exposures and Biomarker Levels
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
Number analyzed (Participants) | 139 | 70
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose until 45 days after last dose of study drug (approximately up to 4 years)
Arm/Group | Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 6.0 mg/kg + Gemcitabine/Docetaxel | Part 1: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel | Part 2: Placebo + Gemcitabine/Docetaxel
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/4 | 8/9 | 76/140 | 35/67
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 6/9 | 106/140 | 45/67
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 9/9 | 140/140 | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel (N=3) | Part 1: MORAb-004 6.0 mg/kg + Gemcitabine/Docetaxel (N=4) | Part 1: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel (N=9) | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel (N=140) | Part 2: Placebo + Gemcitabine/Docetaxel (N=67)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 5 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 2 | 3
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 7 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 8 | 3
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 7 | 6
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MORAb-004 4.0 mg/kg + Gemcitabine/Docetaxel (N=3) | Part 1: MORAb-004 6.0 mg/kg + Gemcitabine/Docetaxel (N=4) | Part 1: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel (N=9) | Part 2: MORAb-004 8.0 mg/kg + Gemcitabine/Docetaxel (N=140) | Part 2: Placebo + Gemcitabine/Docetaxel (N=67)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 8 | 85 | 37
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 8 | 56 | 28
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 32 | 15
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 20 | 11
Lacrimation Increased (Eye disorders) | 0 | 0 | 1 | 8 | 6
Nausea (Gastrointestinal disorders) | 2 | 1 | 5 | 75 | 34
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 54 | 25
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1 | 11 | 15
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 61 | 24
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 38 | 11
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 17 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 10 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 9 | 6
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 8 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 0 | 8 | 4
Fatigue (General disorders) | 3 | 3 | 6 | 103 | 44
Oedema peripheral (General disorders) | 1 | 2 | 2 | 59 | 29
Pyrexia (General disorders) | 2 | 1 | 4 | 51 | 17
Chills (General disorders) | 0 | 1 | 0 | 28 | 3
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 15 | 2
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 12 | 6
Pain (General disorders) | 0 | 0 | 0 | 11 | 4
Asthenia (General disorders) | 0 | 1 | 0 | 7 | 4
Chest Pain (General disorders) | 0 | 0 | 0 | 7 | 2
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 2 | 7 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 17 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 13 | 4
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 9 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 7 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 7 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 7 | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 10 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 3 | 31 | 12
Platelet Count Decreased (Investigations) | 1 | 0 | 0 | 20 | 15
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2 | 16 | 8
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 13 | 7
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 13 | 9
White Blood Cell Count Decreased (Investigations) | 1 | 0 | 0 | 11 | 10
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 10 | 4
Blood Albumin Decreased (Investigations) | 0 | 0 | 0 | 8 | 4
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 8 | 8
Weight Decreased (Investigations) | 0 | 0 | 2 | 8 | 2
Blood Calcium Decreased (Investigations) | 0 | 0 | 0 | 7 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 43 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 19 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 22 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 12 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 8 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 8 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 21 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 25 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 21 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 34 | 13
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 20 | 10
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 14 | 5
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 8 | 2
Headache (Nervous system disorders) | 1 | 2 | 3 | 57 | 13
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 31 | 15
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 16 | 10
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 1 | 16 | 16
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 14 | 7
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 8 | 5
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 24 | 12
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 7 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 42 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 41 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 18 | 10
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 12 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 11 | 5
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 10 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 48 | 21
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 30 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 20 | 3
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 12 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 10 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 10 | 4
Hypertension (Vascular disorders) | 0 | 0 | 0 | 17 | 2
Hot Flush (Vascular disorders) | 0 | 1 | 0 | 9 | 0
Flushing (Vascular disorders) | 1 | 0 | 1 | 7 | 4
Hypotension (Vascular disorders) | 0 | 1 | 0 | 7 | 7
Deafness Unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Catheter Site Rash (General disorders) | 0 | 1 | 0 | 0 | 0
Early Satiety (General disorders) | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Staphylococcal Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other